CLINICAL TRIAL: NCT06857253
Title: A Phase I, Randomized, Double-blind and Dose-escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HRS-1301 Following Single and Multiple Dose Administration in Healthy
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HRS-1301 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-1301-101
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-1301 group (Experimental)
  Interventions: Drug: HRS-1301
- HRS-1301 placebo group (Placebo Comparator)
  Interventions: Drug: HRS-1301 placebo

INTERVENTIONS:
Drug: HRS-1301 — HRS-1301.
  Arms: HRS-1301 group
Drug: HRS-1301 placebo — HRS-1301 placebo.
  Arms: HRS-1301 placebo group

SUMMARY:
This study aims to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of HRS-1301 following single and multiple dose administration in healthy subjects. The study consists of two parts (Part 1 and Part 2) with 82 subjects planned to be enrolled. Possible adjustments to sample size, treatment duration and follow-up time will depend upon emerging data.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects must be at least 18 years old and no more than 55 years old on the date of signing the ICF.
2. The female subjects must be non-pregnant or non-childbearing potential.
3. Subjects must understand the study procedures and methods, voluntarily participate in this study and sign the ICF in person.

Exclusion Criteria:

1. Have a gastrointestinal, liver or kidney disease or other condition known to affect drug absorption, distribution, metabolism and excretion or to reduce adherence, as determined by the investigator.
2. Those who had severe trauma or had undergone surgery within 3 months prior to screening, or planned to undergo surgery during the trial.
3. Have a history of repeated drug allergies.
4. People who have used any drug in the 2 weeks prior to screening.
5. Those who received live (attenuated) vaccine within 4 weeks prior to screening or planned to receive it during the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs) | From the first dose up to Day 21.

SECONDARY OUTCOMES:
HRS-1301 plasma drug concentration. | Up to 168 hours after the first dosing.
HRS-1301 urine drug concentration. | Up to 168 hours after the first dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided